CLINICAL TRIAL: NCT06517394
Title: Open Pilot Trial of a Dyadic Mind-body Program for Cardiac Arrest Survivors and Their Caregivers: Recovering Together After Cardiac Arrest
Brief Title: Open Pilot Trial of a Mind-body Program for Cardiac Arrest Survivors and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexander Presciutti, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001877
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Emotional Distress; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Dyads will participate in 6 30-minute skills-based sessions. Sessions will also include provision of anticipatory guidance and and resources to manage cardiac arrest-specific stressors. A clinical psychologist will deliver all of the sessions. The main intervention goal is to provide dyads with resiliency skills and resources to reduce emotional distress and prevent chronic distress.
  Interventions: Behavioral: Recovering Together after Cardiac Arrest

INTERVENTIONS:
Behavioral: Recovering Together after Cardiac Arrest — The intervention will teach resiliency skills (mindfulness, coping, etc.) to dyads and provider anticipatory guidance and resources to manage stressors specific to cardiac arrest. These sessions will take place in person or on Zoom/telephone, depending on the participant's preference and access to technology.

SUMMARY:
The purpose of this study is to pilot a mind-body intervention for cardiac arrest survivors and their informal caregivers, Recovering Together after Cardiac Arrest. The data the investigators gather in this study will be used to further refine our intervention.

DETAILED DESCRIPTION:
The goal of this study is to refine our proposed intervention Recovering Together after Cardiac Arrest (RT-CA) through an open pilot. The investigators will deliver an open pilot of the intervention (N=5 dyads; 10 participants total) to evaluate initial feasibility and acceptability using exit interviews and pre-post assessments.

The open pilot will take place at Massachusetts General Hospital intensive care units and step-down units. Study clinicians will deliver 6, 30 minute sessions of the intervention (at bedside or on Zoom/telephone, depending on participant preference and access). All participants will complete measures at baseline, and after completion of program (6 weeks). At the completion of the program, participants will engage in an exit interview where they will provide feedback of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Out-of-hospital or in-hospital CA survivor (must have new diagnosis of "cardiac arrest" in electronic medical record from index hospitalization with documented loss of pulse) with an identified caregiver (identified by the survivor who is their primary source of emotional and functional support)
2. Score ≥4 on Short Form of the Mini Mental State Exam
3. Ability and willingness to participate in a hybrid in-person/live video or phone intervention
4. English speaking adults, 18 years or older
5. At least one member of the dyad endorses clinically significant emotional distress during screening (>7 on Hospital Anxiety and Depression Scale subscales)

Exclusion Criteria:

1. Active psychosis, mania, substance dependence, or suicidal intent or plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M Presciutti, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Presciutti AM, La Camera D, Perman SM, Elmer J, Donnino MW, Wu O, Parker RA, Vranceanu AM. Single-arm feasibility trial of a resilience intervention for cardiac arrest survivors and their family caregivers, Recovering Together after Cardiac Arrest. Resuscitation. 2025 Nov;216:110855. doi: 10.1016/j.resuscitation.2025.110855. Epub 2025 Oct 6. PMID 41062056

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 14 (7 dyads enrolled (7 survivors and 7 caregivers for a total of 14 participants).)
Completed | 14 (7 dyads completed (7 survivors and 7 caregivers for a total of 14 participants).)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 14 total participants (7 dyads) participated
Arm/Group | Intervention
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants] — Population: 14 total participants (7 dyads) participated
  Participants
    Survivors: number analyzed (Participants) | 7
    Survivors: <=18 years | 0
    Survivors: Between 18 and 65 years | 3
    Survivors: >=65 years | 4
    Caregivers: number analyzed (Participants) | 7
    Caregivers: <=18 years | 0
    Caregivers: Between 18 and 65 years | 4
    Caregivers: >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 14 total participants (7 dyads) participated
  Participants
    Survivors: number analyzed (Participants) | 7
    Survivors: Female | 4
    Survivors: Male | 3
    Caregivers: number analyzed (Participants) | 7
    Caregivers: Female | 4
    Caregivers: Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 14 total participants (7 dyads) participated
  Participants
    Survivors: number analyzed (Participants) | 7
    Survivors: Hispanic or Latino | 0
    Survivors: Not Hispanic or Latino | 7
    Survivors: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 7
    Caregivers: Hispanic or Latino | 0
    Caregivers: Not Hispanic or Latino | 7
    Caregivers: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 14 total participants (7 dyads) participated
  Participants
    Survivors: number analyzed (Participants) | 7
    Survivors: American Indian or Alaska Native | 0
    Survivors: Asian | 0
    Survivors: Native Hawaiian or Other Pacific Islander | 0
    Survivors: Black or African American | 0
    Survivors: White | 7
    Survivors: More than one race | 0
    Survivors: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 7
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 0
    Caregivers: White | 7
    Caregivers: More than one race | 0
    Caregivers: Unknown or Not Reported | 0
Marital Status [Count of Participants; unit: Participants] — Marital status (married) Population: 14 total participants (7 dyads) participated
  Participants
    Survivors: number analyzed (Participants) | 7
    Survivors | 5
    Caregivers: number analyzed (Participants) | 7
    Caregivers | 5

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility Assessed by the Number of Eligible Dyads Enrolled
Description: Proportion of eligible CA survivor-caregiver dyads that enroll in the intervention amongst those who screen in to the study.
Time Frame: 0 weeks
Population: Analysis population (unit) was the dyad. We analyzed 8 dyads (8 survivors and 8 caregivers or 16 participants total).
Measure: Count of Units; unit: dyads
Units Other Than Participants: dyads
Arm/Group | Intervention
Number analyzed (Participants) | 16
Number analyzed (dyads) | 8
dyads | 7

2. Primary Outcome: Assessment Feasibility Assessed by the Number of Participants With no Measures Missing on All Self-report Questionnaires.
Description: Assessment feasibility was assessed by the number of individual participants (not dyads) that have no measures missing on all self-report questionnaires.
Time Frame: Pre-test (0 weeks) to post-test (6 weeks)
Population: We analyzed 14 individual participants (7 survivors and 7 caregivers) for this benchmark, not dyads.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  Survivors: number analyzed (Participants) | 7
  Survivors | 7
  Caregivers: number analyzed (Participants) | 7
  Caregivers | 7

3. Primary Outcome: Adherence Feasibility Assessed by the Number of CA Survivor-caregiver Dyads Who Begin the Intervention and Complete at Least 4 of 6 Intervention Sessions.
Description: Adherence feasibility was assessed by the number of CA survivor-caregiver dyads who begin the intervention and adhere to it by completing at least 4 of 6 intervention sessions.
Time Frame: Pre-test (0 weeks) to post-test (6 weeks)
Population: We analyzed 7 units (dyads), which is comprised of 14 participants (7 survivors and 7 caregivers).
Measure: Count of Units; unit: dyads
Units Other Than Participants: dyads
Arm/Group | Intervention
Number analyzed (Participants) | 14
Number analyzed (dyads) | 7
dyads | 7

4. Primary Outcome: Therapist Fidelity Assessed by the Proportion of 9 Randomly Selected Sessions in Which the Study Clinician Delivered Fully Delivered All Key Session Content.
Description: Number of sessions in which the therapist adhered 100% to the treatment manual. The study coordinator listened to 9 random RT-CA sessions, and, using a checklist, identified whether the study clinician fully adhered to the content of each session by delivering each key ingredient of the session.
Time Frame: Pre-test (0 weeks) to post-test (6 weeks)
Population: Each unit of analysis was a session recording listened to at random by the research coordinator, which they rated the degree to which the study clinician delivered all key ingredients (rated as fully adherent or not adherent).
Measure: Count of Units; unit: Sessions
Units Other Than Participants: Sessions
Arm/Group | Intervention
Number analyzed (Participants) | 9
Number analyzed (Sessions) | 9
Sessions | 7

5. Primary Outcome: Number of Participants With Client Satisfaction Score Greater Than the Midpoint (7.5).
Description: The proportion of participants that scored above the midpoint on the Client Satisfaction Questionnaire-3 (CSQ-3), which assesses satisfaction with a program. Total scores range from 3-12 (midpoint 7.5); higher scores indicate greater satisfaction.
Time Frame: Post-test (6 weeks)
Population: Analysis population was number of participants that scores above the midpoint on the CSQ-3, not dyads.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants | 14

6. Primary Outcome: Credibility and Expectancy Assessed by the Number of Individuals That Score Above the Midpoint on Each Sub-scale of the Credibility and Expectancy Questionnaire
Description: Number of individuals that score above the midpoint on each sub-scale of the Credibility and Expectancy Questionnaire (CEQ). Through two subscales, the CEQ assesses participants' perceptions that a program is logical (credible) and their expectancy that participation would lead to improvements (expectancy). Scores on the credibility subscale range from 3-27 (midpoint 15) and scores on the expectancy factor range from 3-31 (midpoint 17); higher scores on each indicate greater credibility and expectancy.
Time Frame: Pre-test (0 weeks)
Population: For credibility and expectancy, we analyzed individual participant responses on each sub scale (Credibility and expectancy).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  Survivors that endorsed credibility: number analyzed (Participants) | 7
  Survivors that endorsed credibility | 7
  Caregivers that endorsed credibility: number analyzed (Participants) | 7
  Caregivers that endorsed credibility | 4
  Survivors that endorsed expectancy: number analyzed (Participants) | 7
  Survivors that endorsed expectancy | 6
  Caregivers that endorsed expectancy: number analyzed (Participants) | 7
  Caregivers that endorsed expectancy | 1

7. Secondary Outcome: Mean Change in the Hospital Depression and Anxiety Scale Total Score.
Description: Assesses emotional distress in medical patients; total scale ranges from 0-42, higher scores represent worse distress. A negative mean change in the total score means emotional distress improved.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: Analyzed change in total score in individual survivors and caregivers
Measure: Mean (95% Confidence Interval); unit: mean change units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
mean change units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | -10.6 [-14.6 to -6.6]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | -6.6 [-11.2 to -1.9]

8. Secondary Outcome: Mean Change in Post-Traumatic Stress Disorder Checklist - 5 Total Score.
Description: 20-item questionnaire that measures post-traumatic stress disorder symptoms. Scores range from 0 to 80, with higher scores indicating greater severity and intensity of symptoms. A negative change in the total score represents improvement in symptoms.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: Analyzed change in 7 survivors and 7 caregivers
Measure: Mean (95% Confidence Interval); unit: mean change units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
mean change units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | -17.6 [-34 to -1.1]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | -6.3 [-11 to -1.6]

9. Secondary Outcome: Mean Change in The Cognitive and Affective Mindfulness Scale-Revised Total Score
Description: Measures dispositional mindfulness, total scores range from 12-48, higher values reflect higher levels of mindfulness. A positive mean change in the total score reflected increased dispositional mindfulness.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: Analyzed change in 7 survivors and 7 caregivers
Measure: Mean (95% Confidence Interval); unit: mean change units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
mean change units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | 5.4 [0.4 to 10.4]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | 1.5 [-2.5 to 5.4]

10. Secondary Outcome: Mean Change in Enhancing Recovery in Coronary Heart Disease Social Support Inventory Total Score
Description: 7-item measure that assesses perceived social support. Higher scores indicate greater social support. Total scores range from 8 to 34. A positive mean change in the total score indicates increases in perceived social support.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: Analyzed change in 7 survivors and 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | 1.9 [-1 to 4.8]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | 0 [-3.7 to 3.7]

11. Secondary Outcome: Mean Change in Measure of Current Status Part A (MOCS-A) Average Score.
Description: Assesses ability to engage in a series of healthy coping skills (e.g., relaxation, social support, adaptive thinking). Higher scores indicate a stronger ability to recognize stress and cope. Scores are averaged and range from 0-4. A positive change in the MOCS-A average score indicates improvements in coping.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: Analyzed change in 7 survivors and 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  survivors: number analyzed (Participants) | 7
  survivors | 0.3 [-0.3 to 0.9]
  caregivers: number analyzed (Participants) | 7
  caregivers | 0.2 [-0.4 to 0.9]

12. Secondary Outcome: Mean Change in the World Health Organization Quality of Life-Brief Sub Scale Scores
Description: 26-item measure assessing quality of life across four domains: physical health, psychological health, social relationships, and environment. Higher scores indicate higher quality of life for all domains. Scores in each domain range from 4 to 20. Scores were assessed at pre- and post-test; a positive mean change score in each domain indicates improved quality f life.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: 7 survivors and 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  survivors phys QOL: number analyzed (Participants) | 7
  survivors phys QOL | 2.2 [-0.9 to 5.3]
  caregivers phys QOL: number analyzed (Participants) | 7
  caregivers phys QOL | -0.08 [-0.5 to 0.4]
  survivors psych QOL: number analyzed (Participants) | 7
  survivors psych QOL | 1 [-0.3 to 2.4]
  caregivers psych QOL: number analyzed (Participants) | 7
  caregivers psych QOL | 0.5 [-0.5 to 1.5]
  survivors soc QOL: number analyzed (Participants) | 7
  survivors soc QOL | 1 [-1.4 to 3.3]
  caregivers soc QOL: number analyzed (Participants) | 7
  caregivers soc QOL | -0.4 [-1.6 to 0.8]
  survivors env QOL: number analyzed (Participants) | 7
  survivors env QOL | -0.4 [-1.3 to 0.5]
  caregivers env QOL: number analyzed (Participants) | 7
  caregivers env QOL | -0.07 [-1.1 to 0.9]

13. Secondary Outcome: Mean Change in Dyadic Relationship Scale Sub Scales
Description: Questionnaire that assesses perceptions of dyadic interactions from both members of the relationship. The caregiver version is 11 items and the patient version is 10 items. Scores are calculated for two subscales: dyadic strain (scores range from 0-15) and positive interactions (scores range from 0-18). Lower scores on the dyadic strain subscale and greater scores on the positive interactions subscale indicate fewer relationship stressors and more positive aspects of the relationship.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: 7 survivors 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  survivors positive: number analyzed (Participants) | 7
  survivors positive | 0 [-5.1 to 5.1]
  caregivers positive: number analyzed (Participants) | 7
  caregivers positive | 0.3 [-1.2 to 1.8]
  survivors strain: number analyzed (Participants) | 7
  survivors strain | 0.1 [-4 to 3.7]
  caregivers strain: number analyzed (Participants) | 7
  caregivers strain | 0.7 [-1.1 to 2.5]

14. Secondary Outcome: Mean Change in Dyadic Coping Inventory Sub Scales
Description: Measures perceived quality of dyad's communication and proficiency in using adaptive dyadic coping skills. Subscales are summed for a total subscale score. Higher scores indicate greater quality communication and/or coping.
  Stress communicated by oneself measures how well stress is communicated by oneself to their partner Range 4-20.
  Stress communicated by one's partner Measures how well one's partner communicates about their stress. Range 4-20.
  Supportive coping provided by one's partner Measures the quality of emotional and/or problem-focused support provided by one's partner Range 5-25.
  Negative dyadic coping by one's partner Measures the degree that one's partner uses hostile, ambivalent, and superficial actions/words that have deleterious intentions. Range 4-20.
  Joint or common coping Measures the degree to which dyads work together to manage stress.Range 5-25.
  Evaluation of dyadic coping Measures perception of the quality of the dyad's approach to coping.Range 2-10.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: Analyzed change in 7 survivors and 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  Survivors stress communicated by oneself: number analyzed (Participants) | 7
  Survivors stress communicated by oneself | 0 [-3.5 to 3.5]
  Caregivers stress communicated by oneself: number analyzed (Participants) | 7
  Caregivers stress communicated by oneself | 2.6 [0 to 5.2]
  Survivors stress communicated by partner: number analyzed (Participants) | 7
  Survivors stress communicated by partner | 1.9 [-1.2 to 4.9]
  Caregivers stress communicated by partner: number analyzed (Participants) | 7
  Caregivers stress communicated by partner | 0.8 [-1.6 to 3.3]
  Survivors supportive coping provided by partner: number analyzed (Participants) | 7
  Survivors supportive coping provided by partner | 2.2 [-3.1 to 7.4]
  Caregivers supportive coping provided by partner: number analyzed (Participants) | 7
  Caregivers supportive coping provided by partner | 1.9 [-3.9 to 7.6]
  Survivors negative dyadic coping by partner: number analyzed (Participants) | 7
  Survivors negative dyadic coping by partner | 2.2 [0.2 to 4.1]
  Caregivers negative dyadic coping by partner: number analyzed (Participants) | 7
  Caregivers negative dyadic coping by partner | 1.8 [-2.5 to 6.2]
  Survivors common dyadic coping: number analyzed (Participants) | 7
  Survivors common dyadic coping | 1 [-4 to 6]
  Caregivers common dyadic coping: number analyzed (Participants) | 7
  Caregivers common dyadic coping | 0.9 [-2.5 to 4.2]
  Survivors evaluation of dyadic coping: number analyzed (Participants) | 7
  Survivors evaluation of dyadic coping | 0.9 [-3.1 to 7.4]
  Caregivers evaluation of dyadic coping: number analyzed (Participants) | 7
  Caregivers evaluation of dyadic coping | 0.4 [-1.9 to 2.7]

15. Secondary Outcome: Mean Change in Applied Mindfulness Scale Total Score.
Description: 15-item questionnaire measuring how participants use mindfulness when facing stressors. Scores range from 0 to 60 with higher scores indicating greater use of mindfulness practices.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: 7 survivors 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | -2.5 [-11.9 to 7.1]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | 2.7 [-3.7 to 9.2]

16. Secondary Outcome: Mean Change in Preparedness for Caregiving Scale Total Score
Description: For caregivers, this scale measures caregiver preparedness to care for survivor. In this study, for survivor participants, we adapted the language to measure preparedness to care for oneself. Scores range from 0 to 32 Higher scores indicate greater perceived readiness for caregiving (for caregivers) or for survivorship (for survivors).
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: 7 survivors 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | 5.4 [-1.6 to 12]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | 3.1 [-3.5 to 9.7]

17. Secondary Outcome: Mean Change in Meaning in Life Questionnaire Sub Scales
Description: 10 items measuring presence of meaning and purpose in life. Assesses two dimensions: presence and search. Items are rated on a 7-point scale from 1 (Absolutely Untrue) to 7 (Absolutely True). Both presence of meaning and search for meaning subscale scores range from 5-35. Higher scores indicate greater presence and search.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: 7 survivors 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  Survivors presence: number analyzed (Participants) | 7
  Survivors presence | -2.2 [-5.6 to 1.1]
  Caregivers presence: number analyzed (Participants) | 7
  Caregivers presence | 0.2 [-3.2 to 3.4]
  Survivors search: number analyzed (Participants) | 7
  Survivors search | -5 [-13.9 to 4]
  Caregivers search: number analyzed (Participants) | 7
  Caregivers search | 0.5 [-2.4 to 3.5]

18. Secondary Outcome: Gratitude Questionnaire Six Item Form
Description: Measures participant's gratitude disposition. Each item is rated on a 7-point Likert scale. Scores range from 6 to 42. Higher scores indicate a more grateful disposition.
Time Frame: Pre-test (0 weeks), Post-Test (6 weeks)
Population: 7 survivors 7 caregivers
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 14
change in units on a scale
  Survivors: number analyzed (Participants) | 7
  Survivors | -0.9 [-2.6 to 0.9]
  Caregivers: number analyzed (Participants) | 7
  Caregivers | 0 [-3.7 to 3.7]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Intervention: Survivors: This arm represents the survivors that participated in the intervention.
  Dyads of cardiac arrest survivors and their caregivers participated in 6 30-minute skills-based sessions. Sessions included provision of anticipatory guidance and and resources to manage cardiac arrest-specific stressors. A clinical psychologist delivered all of the sessions. The main intervention goal was to provide dyads with resiliency skills and resources to reduce emotional distress and prevent chronic distress.
  Recovering Together after Cardiac Arrest: The intervention taught resiliency skills (mindfulness, coping, etc.) to dyads and provider anticipatory guidance and resources to manage stressors specific to cardiac arrest. These sessions took place in person or on Zoom/telephone, depending on the participant's preference and access to technology.
- Intervention: Caregivers: This arm represents the caregivers that participated in the intervention.
  Dyads of cardiac arrest survivors and their caregivers participated in 6 30-minute skills-based sessions. Sessions included provision of anticipatory guidance and and resources to manage cardiac arrest-specific stressors. A clinical psychologist delivered all of the sessions. The main intervention goal was to provide dyads with resiliency skills and resources to reduce emotional distress and prevent chronic distress.
  Recovering Together after Cardiac Arrest: The intervention taught resiliency skills (mindfulness, coping, etc.) to dyads and provider anticipatory guidance and resources to manage stressors specific to cardiac arrest. These sessions took place in person or on Zoom/telephone, depending on the participant's preference and access to technology.
Arm/Group | Intervention: Survivors | Intervention: Caregivers
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT06517394/Prot_SAP_000.pdf